CLINICAL TRIAL: NCT02673333
Title: A Phase II Clinical Trial of Single Agent Pembrolizumab in Subjects With Advanced Adrenocortical Carcinoma
Brief Title: Single Agent Pembrolizumab in Subjects With Advanced Adrenocortical Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-286
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Results first posted 2020-01-06 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Adrenocortical Carcinoma
Keywords: Pembrolizumab; 15-286
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — pembrolizumab

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab 200 mg will be administered as a 30 minute IV infusion Q3W.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab

SUMMARY:
Pembrolizumab is a type of immunotherapy, and the purpose of this study is to find out what effects, good and/or bad, pembrolizumab has on you, and your cancer.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Be ≥ 18 years of age on day of signing informed consent.
* Have histologically- or cytologically- confirmed unresectable or metastatic ACC that is considered incurable by local therapies.
* Have an ECOG performance status of 0 or 1.
* Have measurable disease based on RECIST v1.1
* Have provided tissue for PD-L1 biomarker analysis from either archived tissue or a newly obtained core or excisional biopsy.
* Consent for use of archived tissue for research purposes.
* Demonstrate adequate organ function, all screening labs should be performed within 28 days of treatment initiation.

Hematological

* Absolute neutrophil count (ANC) ≥1,500 /mcL
* Platelets ≥100,000 / mcL Renal
* Serum creatinine ≤1.5 X upper limit of normal (ULN) OR Measured or calculateda creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN Hepatic
* Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
* AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases Coagulation
* International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants aCreatinine clearance should be calculated per institutional standard.

  * Female subjects of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
  * Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free of menses for >1 year.
  * Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks prior to the first dose of trial treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. The use of physiologic doses of corticosteroids for adrenal and pituitary insufficiency is not considered a form of systemic steroid therapy and would not exclude a subject from the study.
* Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

  °Note: Subjects with ≤ Grade 2 neuropathy or ≤ Grade 2 alopecia are an exception to this criterion and may qualify for the study.
* If subject underwent major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Has known active central nervous system metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for brain metastases for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study. Subjects that have adrenal or pituitary insufficiency that require physiologic corticosteroid replacement therapy would not be excluded from the study.
* Has evidence of interstitial lung disease or history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.

Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-02; Primary Completion 2019-01-11 (Actual); Study Completion 2026-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nitya Raj, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - University of Michigan (Data or Specimen Analysis Only), Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Raj N, Zheng Y, Kelly V, Katz SS, Chou J, Do RKG, Capanu M, Zamarin D, Saltz LB, Ariyan CE, Untch BR, O'Reilly EM, Gopalan A, Berger MF, Olino K, Segal NH, Reidy-Lagunes DL. PD-1 Blockade in Advanced Adrenocortical Carcinoma. J Clin Oncol. 2020 Jan 1;38(1):71-80. doi: 10.1200/JCO.19.01586. Epub 2019 Oct 23. PMID 31644329
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab: Pembrolizumab 200 mg will be administered as a 30 minute IV infusion Q3W.
  Pembrolizumab
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 62 [19 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 36
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: using RECIST v1.1 A Simon two stage minimax design will be employed to carry out this objective. In the first stage, 21 patients will be enrolled. If at least 3 out of 21 patients respond (partial response - PR or complete response - CR), we will enroll an additional 18 patients for a total of 39 patients. At the end of the study, 8 of 39 patients will need to respond to consider the therapy promising. The study will be complete when all subjects have either completed 24 months of drug therapy, progressed, or discontinued from the study for other reasons.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 39
Participants
  Complete Response | 0
  Partial Response | 9
  Stable Disease | 7
  Progressive Disease | 15
  Could Not Be Evaluated | 8

ADVERSE EVENTS:
Time Frame: Up to 24 months
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 20/39
Serious Adverse Events (participants affected / at risk) | 5/39
Other Adverse Events (participants affected / at risk) | 23/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=39)
Increased AST/ALT (Investigations) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=39)
Increased AST/ALT (Investigations) | 9
Hypocalcemia (Metabolism and nutrition disorders) | 4
Increased Alkaline Phosphatase (Investigations) | 4
Lymphopenia (Investigations) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Increased Creatinine (Investigations) | 2
Fatigue (General disorders) | 8
Chills (General disorders) | 2
Hypothyroidism (Endocrine disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 3
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/33/NCT02673333/Prot_SAP_000.pdf